CLINICAL TRIAL: NCT04092803
Title: Virtual Reality as a Distraction Technique for Performing Lumbar Punctures in Children and Young Adults With Leukemia: a Feasibility Study
Brief Title: Virtual Reality as a Distraction Technique for Performing Lumbar Punctures in Children and Young Adu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-0994.cc; P30CA046934 (NIH)
Record Dates: First submitted 2019-06-11; First posted 2019-09-17 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA for LP (No Intervention): Patients who decline to undergo an LP with VR will be asked if they would be willing to participate by answering questionnaires specific to their pre procedure anxiety. This will include questionnaires 2 and 3 from above. The investigators will also plan to collect vital sign data if they agree to participate in that capacity.
- VR for LP (Experimental): The patients in this study will be presented the opportunity to use VR instead of undergo GA for a LP. Patients who agree to undergo an LP with VR will be assessed by a certified child life specialist (CCLS) to determine whether the patient is an appropriate candidate for using VR.The system includes a VR headset with VR software already loaded in to it. The VR software to be used is either a game called "Pebbles the Penguin" or "SpacePups" (Weightless Studios).
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — The system includes a VR headset with VR software already loaded in to it.
  Arms: VR for LP

SUMMARY:
The goal of this feasibility study is to determine if Virtual Reality (VR) can be adequately used as an alternative to General Anesthesia (GA) for Lumbar Punctures (LP).

DETAILED DESCRIPTION:
The primary purpose of this study is to determine the feasibility of implementing VR as an alternative to general anesthesia in adolescents and young adults with leukemia who undergo LPs for maintenance of chemotherapy. The patients in this study will be presented the opportunity to use VR instead of undergo GA for a LP. Success will be defined as successful performance of the procedure with VR instead of GA.

Additionally, we plan to administer questionnaires to all patients approached for the trial if they are willing, even if they decide not to use VR for their LP. These questionnaires are listed below.

Studies have linked the use of technology with decreased distress, increased cooperation, and improved pain management. For example, pediatric patients who had access to a video game to engage for distraction during anesthesia induction for surgery were less distressed and more cooperative during mask induction. In children and adolescents requiring port access VR distraction was significantly better than standard of care in terms of reducing physiological arousal (i.e., pulse rate) and pain ratings. VR has been utilized effectively in the management of pediatric and adult wound care, burn care, and dressing changes. Patients who had dressing changes while immersed in VR used less pain medication, had lower pain scores and often requested to use VR for future dressing changes all while having their procedures take less time. Simple distraction techniques might not be enough. One study evaluated the effectiveness of using augmented reality with children undergoing burn dressing changes. They compared augmented reality to standard distraction with an age appropriate video game. The study found augmented reality reduced pain scores significantly better than video game distraction.

When not accompanied by appropriate pain control, stressful and invasive medical procedures can lead to posttraumatic stress symptoms and negative reactions or noncompliance to subsequent medical experiences. Specifically, adults who experienced more medical fear and pain as children were more likely to rate their adult medical fear and pain higher and avoid medical care. Pharmacological strategies alone are often not enough to effectively manage a child's pain. Non-pharmacological pain management uses alternative strategies, such as distraction, to replace or augment medication to help reduce a child's pain. VR systems have been successfully trialed in a small number of patients, mostly adolescents and adults. VR has reliably demonstrated decreased pain, anxiety, suffering, time spent thinking about pain and perceived time spent in a medical procedure.

Typically, VR has to be experienced seated upright or standing with few exceptions because of the design of the software. Patients underoing LP are often required to lay laterally, as is the case with this study. Therefore, we will be using VR software (Pebbles the Penguin and SpacePups, Weightless Studios) that is age appropriate for the study population, engaging enough for young adults, and designed to be reoriented to the patient's position.

The goal of this feasibility study is to determine if VR can be adequately used as an alternative to GA for LP. Utilizing distraction will eliminate the risk associated with general anesthesia, and the accompanying inconvenience of general anesthetic exposure on these patients perioperatively, as well as long term. Additionally, we wish to decrease the burden of cost for these procedures as currently practiced. LPs performed under GA require the presence of an anesthesiologist, medications, and recovery staff, all of which add increased cost to the procedure. With this VR system, there is a one time cost associated with the purchase of the system (in our case, the VR system was donated to our hospital by a non-profit called The Starlight Foundation), and the system can be used multiple times on multiple patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric and young adult patients 10-25 years of age
2. Lumbar puncture for chemotherapy per leukemia therapy
3. Cognitively appropriate
4. Assessed by child life specialist as appropriate to use VR
5. Previous LP with GA
6. Tested negative for COVID-19

Exclusion Criteria:

1. History of seizures
2. Active headache
3. Active nausea or vomiting
4. ASA (American Society of Anesthesiologists) greater than 4
5. Allergy to lidocaine, procaine, or propofol
6. Developmental delay
7. No previous LP with GA
8. Tested positive for COVID-19, or opted out of of COVID-19 testing

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Success of completion of the LP with VR | 4 months
  This is a feasibility study with the primary outcome defined as success of completion of the Lumbar Puncture with Virtual Reality.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (Pain VAS) | 4 months
  This is a numerical scale from 0 to 10, 0 being no pain, 10 being the worst possible pain.
Child Anxiety Meter-State (CAM-S) | 4 months
  The CAM-S is a vertical analog scale for child self-report of state anxiety. Children are asked to rate how nervous or worried they feel "right now" by marking a line on a visual depiction of a thermometer. Lines closet to the bottom of the thermometer indicate less worry, while lines towards the top of the thermometer indicate more worry. The scale ranges from Calm (score of 0) to very very nervous (score of 100)
Children's Fear Scale (CFS) | 4 months
  The Children's fear Scale is a one-item scale that consists of a row of faces with expressions ranging from no fear (score of 0) to extreme fear (score of 4). Children are asked to choose the face that most closely reflects how anxious or fearful they are feeling.

CONTACTS AND LOCATIONS:
Overall Officials: James Thomas, MD, Principal Investigator — Physician
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No